CLINICAL TRIAL: NCT01027039
Title: The Effect of Mozart Music on Visual Field Testing in Glaucoma Patients: Will Music Tame the Savage Perimeter?
Brief Title: Will Listening to Music Make it Easier to Take a Visual Field Test?
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jonathon Myers, Attending Surgeon, Wills Eye
Other Study IDs: 07-829E
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: primary open angle glaucoma; pigmentary glaucoma; exfoliative glaucoma; angle closure glaucoma; low tension glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients using noise-reducing headphones: Patients using noise-reducing headphones
- Patients using no headphones: Patients using no headphones
- Patients using headphones with music: Patients using headphones with music

SUMMARY:
The purpose of this study is to examine if there is a difference between glaucoma patients having background music and not having background music before visual field testing.

DETAILED DESCRIPTION:
Glaucoma is one of the leading causes of blindness in the United States. Over 2.5 million people in the United States have glaucoma. The goal of ophthalmologists is two-fold: 1) to detect glaucoma early, and 2) to stop the progression of disease and subsequent visual loss.

Many parameters are used to detect and follow glaucoma over the patient's lifetime including optic nerve appearance, intraocular pressure by applanation and visual field perimetry testing results. Perimetry testing aims to detect visual field loss that may be associated with glaucoma and institute more aggressive treatment measures when necessary. However, it is suspected that 50% or more of the optic nerve fibers are already irreversibly damaged before a visual field defect can be identified on testing. Furthermore, the patient's ability to take a visual field test is paramount in the doctor's ability to interpret the test. That is, if a visual field test taker performs the test with low reliability (i.e. too many false positive, false negative or fixation losses), the interpretability of the test by the ophthalmologist is difficult or impossible.

Interestingly, a recent study in the British Journal of Ophthalmology suggested the positive effect Mozart music has on visual field test taking ability. This study showed better first time automated perimetry performance in normals immediately following exposure to the first 10 minutes of Mozart's Sonata for Two Pianos in D Major. The music group had 20 times fewer fixation losses, three times fewer false positive responses and 10 times fewer false negative responses.

No study has determined if Mozart music improves the reliability indices of Humphrey visual field testing for glaucoma patients or experienced test takers. In efforts to improve patient's reliability on visual field testing, we propose a randomized controlled trial to determine if listening to music before field testing improves testing reliability.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 40-80 years
* Best corrected visual acuity: 20/50 or better in both eyes
* Experienced visual field test takers only: Patient has taken at least 2 prior visual field tests
* Mean defect values: MD no greater than 15
* Reliability on prior visual field indices must each be less than or equal to 40%
* Glaucoma type: Open angle glaucoma (including primary open angle glaucoma, pigmentary glaucoma and exfoliative glaucoma) angle closure glaucoma and low tension glaucoma
* Visual field testing program: Humphrey 24-2 Sita Standard
* Number of eyes per patient: Both (2) eyes will be tested for each subject

Exclusion Criteria:

* Patients with other ocular disease affecting central vision other than mild- moderate nuclear sclerosis (i.e. patients with macular scar, age-related macular degeneration, diabetic retinopathy, etc.)
* Systemic conditions affecting ability to take HVF (i.e. dementia, CVA, severe arthritis, etc.)
* Any visual field taken that is not the Humphrey 24-2 SITA Standard field will not be acceptable

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma service
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Myers, Principal Investigator — Wills Eye
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript has been published.

REFERENCES:
- [Background] Shue B, Chatterjee A, Fudemberg S, Katz LJ, Moster MR, Navarro MJ, Pro M, Schmidt C, Spaeth GL, Stirbu O, Yalcin A, Myers JS. The effects of Mozart's music on the performance of glaucoma patients on automated perimetry. Invest Ophthalmol Vis Sci. 2011 Sep 21;52(10):7347-9. doi: 10.1167/iovs.11-7430. PMID 21828156